CLINICAL TRIAL: NCT06015269
Title: Exploratory Study on Baize DC Injection in Preventing Recurrence and Metastasis After Radical Tumor Surgery
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Cell Therapy Group Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BZT003-A-01
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumor
Keywords: Solid tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DC cells (Experimental): Super DC Vaccine (DC)
  Interventions: Drug: DC cells

INTERVENTIONS:
Drug: DC cells — At a single arm, 1x107cells dose
  Other Names: Super DC Vaccine (DC)

SUMMARY:
This is an exploratory study on the safety, immune response, and preliminary effectiveness of single arm, fixed dose therapy

DETAILED DESCRIPTION:
This study is a clinical study exploring the safety, immune response, and preliminary efficacy of a single arm, 1x107cells dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old, weight ≥ 40kg; No gender limit;
2. Subjects with malignant solid tumors diagnosed by histology or cytology and undergoing radical resection surgery;
3. At the beginning of the study (after surgery), there were no lesions, no local recurrence or distant metastasis on the imaging, and no brain metastasis (images within one month before enrollment can be used for screening);
4. Subjects in the safety verification stage need to provide immunohistochemical test results with positive expression of Survivin or P53;
5. ECOG score 0-1 points;
6. There are sufficient venous channels and no contraindications for peripheral blood mononuclear cell collection surgery;
7. Organs and bone marrow function well:

   1. Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50% evaluated by echocardiography within one month of enrollment; The electrocardiogram is basically normal;
   2. Platelets ≥ 90 × 10 ^ 9/L;
   3. Hemoglobin ≥ 90g/L (no blood transfusion or erythropoietin dependence within 7 days);
   4. Total bilirubin ≤ 2 times the upper limit of normal value;
   5. Serum creatinine ≤ 1.5 times the upper limit of normal value;
   6. Transaminases (AST, ALT) ≤ 2.5 times the upper limit of normal value (if liver cancer is 5 times the upper limit of normal value);
   7. International standardized ratio (INR) or prothrombin time (PT) ≤ 1.5 times the upper limit of normal value;
   8. Pulmonary function: ≤ CTCAE level 1 dyspnea and SaO2 ≥ 91% in indoor air environment;
8. Able to understand trial requirements and matters, willing to participate in clinical research according to trial requirements;

Exclusion Criteria:

1. HIV and syphilis serological reactions were positive; Hepatitis B surface antigen is positive, hepatitis B core antibody is positive, and the copy number of hepatitis B virus DNA is higher than the lower limit of detection and or greater than or equal to 1000 copies/ml; Or hepatitis C virus infected individuals;
2. Any uncontrollable active infection, coagulation disorder, or any other major disease;
3. Pregnant or lactating women
4. Suffering from active neuroautoimmune or inflammatory diseases, such as any of the following: inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, multiple sclerosis, Sjogren's syndrome, etc., and receiving relevant treatment; Subjects who are still using immunosuppressants for organ transplantation; Or subjects who have been using immunosuppressive drugs such as glucocorticoids for a long time cannot stop at least 4 weeks before enrollment; Severe allergic constitution;
5. Subjects with existing abnormalities in the central nervous system, such as seizures, cerebral vascular ischemia/bleeding, dementia, cerebellar diseases, or any autoimmune diseases associated with central nervous system involvement;
6. Major cardiovascular diseases with clinical significance include:

   Symptomatic congestive heart failure

   B Unstable angina pectoris

   Severe arrhythmia requiring medication treatment

   Uncontrolled hypertension

   Myocardial infarction or ventricular arrhythmia within 6 months prior to screening
7. Other situations where researchers believe it is not suitable to participate in clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | within 1 months of single injection
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Lou jinxing, Principal Investigator — Shanghai Mengchao Cancer Hospital
Locations (1):
- Shanghai Mengchao Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR